CLINICAL TRIAL: NCT02392104
Title: Prospective Evaluation of an Extended Interval of INR Follow-up in a VA Anticoagulation Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William S. Middleton Memorial Veterans Hospital (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Carla Staresinic, Manager, Anticoagulation Services, William S. Middleton Memorial Veterans Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1296
Record Dates: First submitted 2015-02-25; First posted 2015-03-18 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Anticoagulation
Keywords: International Normalized Ratio; Warfarin
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental): All patients in the study will be in the intervention arm.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — If the patient's INRs stay within goal range, their interval of INR follow-up will be extended based on a protocol to a maximum of 12 weeks.
  Other Names: Coumadin

SUMMARY:
The purpose of this study is to determine the feasibility, safety, and acceptability of implementing an extended interval of INR follow-up in Veterans on a stable dose of warfarin in the Anticoagulation Clinic at the William S. Middleton Memorial Veterans Hospital.

All participants will be provided usual care from the anticoagulation clinic, except for the interval between INRs. If the participant continues to be on a stable dose of warfarin and the INRs are within the goal range of 2-3 (including lab variation), follow-up visits will be scheduled following an extended interval protocol. Patient satisfaction will be evaluated at various points throughout the study. Additionally provider satisfaction, confidence, and knowledge of the extended interval protocol will be analyzed. Bleeding and thromboembolic events will be evaluated to ensure the safety of an extended follow-up interval.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility, safety, and acceptability of implementing an extended interval of INR follow-up in Veterans on a stable dose of warfarin in the Anticoagulation Clinic at the William S. Middleton Memorial Veterans Hospital.

All participants will be provided usual care from the anticoagulation clinic, except for the interval between INRs. If the participant continues to be on a stable dose of warfarin and the INRs are within the goal range of 2-3 (including lab variation), follow-up visits will be scheduled following an extended interval protocol, from 5-6 weeks, to 7-8 weeks, to 11-12 weeks and then continued with 11-12 week visits if INRs continue to remain in goal range and appropriate for the patient. Patient satisfaction will be evaluated at baseline, 6-, 12-, and 24-months. Additionally provider satisfaction, confidence, and knowledge of the extended interval protocol will be analyzed. Bleeding and thromboembolic events will be evaluated to ensure the safety of an extended follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* requirement for indefinite warfarin therapy
* target INR of 2-3
* stable weekly warfarin dose for the past 6 months (not more than a single, one-time adjustment (boost/omission) in the past 6 months, planned interruption for a procedure or surgery with INR(s) out of range in the past 6 months would not exclude a patient)
* a patient of the Madison VA anticoagulation clinic for the previous 12 months

Exclusion Criteria:

* consistently drink ≥4 alcoholic beverages/day or a documented episode of alcohol binging in the past 6 months
* diagnosis of cancer and on active chemotherapy/radiotherapy in the past 3 months
* life expectancy of < 1 year
* enrolled in other investigational drug protocols
* only receiving anticoagulation care at the Madison VA for part of the year (e.g. snowbirds)
* receiving visiting nurse services for INR monitoring
* thrombocytopenia (<100K) within past 12 months
* history of bleeding or thromboembolism requiring medical intervention within past 6 months
* treatment for active liver disease (e.g. hepatitis)
* diagnosis or documentation in EMR suggesting cognitive impairment
* activated power of attorney
* inability to provide informed consent
* non-English speaking
* unstable mental health disorder that impairs judgment
* history of non-adherence to anticoagulation clinic policies and procedures (i.e. missed appointments, self-adjustment of warfarin dose, nonadherence, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Staresinic, PharmD, Principal Investigator — William S. Middleton Memorial Veterans Hospital

REFERENCES:
- [Derived] Schoen RR, Nagy MW, Porter AL, Margolis AR. Patient Satisfaction With Extended International Normalized Ratio Follow-up Intervals in a Veteran Population. Ann Pharmacother. 2020 May;54(5):442-449. doi: 10.1177/1060028019889414. Epub 2019 Nov 21. PMID 31752504

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended INR Follow-up Interval Group: All patients in the study will be in the intervention arm.
  Warfarin: If the patient's INRs stay within goal range, their interval of INR follow-up will be extended based on a protocol to a maximum of 12 weeks.
Period: Overall Study
Arm/Group | Extended INR Follow-up Interval Group
Started | 50 (one participant enrolled but was removed prior to starting study protocol)
Completed | 39
Not Completed | 11
Not completed — discontinuation of warfarin | 3
Not completed — bleeding event | 1
Not completed — transferred care to another doctor | 2
Not completed — INR goal range changed | 1
Not completed — admitted to skilled nursing facility | 3
Not completed — INRs drawn by visiting nurse services | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 50
HAS-BLED score [Mean (Standard Deviation); unit: units on a scale] — The HAS-BLED score evaluates a patient's bleeding risk. HAS-BLED is the official name of the tool to assess risk. Scores range from 0-9. Scores of 3 or higher indicate a high bleeding risk.
  units on a scale | 1.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Participant Accrual
Description: Number of participants who enroll vs. number of individuals invited
Time Frame: up to 2.25 years
Population: 107 invited to participate in the study, not all enrolled or started the study
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 107
Participants
  Number of patients invted | 107
  Patient enrolled in study | 51
  Patients analyzed for study | 50

2. Primary Outcome: Number of Participants Able to be Scheduled for at Least One 12-week Interval
Description: This outcome will determine the number of participants able to be scheduled for at least one 12-week interval
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 50
Participants | 36

3. Primary Outcome: Number of Participants Scheduled for at Least 4 Consecutive 12-week Intervals
Description: The outcome will determine the number of participants scheduled for at least 4 consecutive 12-week intervals
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 50
Participants | 15

4. Secondary Outcome: Change in Frequency of Appointments From Baseline to End of Study
Description: This outcome will evaluate the change in frequency of appointments from baseline to end of study (at 12 and 24 months)
Time Frame: 12 and 24 months
Population: 44 participants remained in the study at 12 months
Measure: Mean (Standard Deviation); unit: visits per 12 months
Arm/Group | Intervention Arm
Number analyzed (Participants) | 44
visits per 12 months
  Planned anticoagulation visits (baseline) | 12.67 (2.56)
  Planned anticoagulation visits (0-12 months) | 10.43 (3.58)

5. Secondary Outcome: Bleeding and Thromboembolic Events From Baseline
Description: This outcome will determine the number of bleeding and thromboembolic events from baseline
Time Frame: 24 months
Measure: Number; unit: events
Arm/Group | Intervention Arm
Number analyzed (Participants) | 50
events
  Number of thromboembolic events | 2
  Number of major bleeding events | 6
  Number of serious bleeding events | 16

6. Secondary Outcome: Change in Time in Therapeutic Range From Baseline
Description: The outcome will evaluate the change in time in therapeutic range (TTR) from baseline (intention-to-treat)
Time Frame: 6, 12, and 24 months
Population: 49 participants at 12 months, 44 participants at 24 months
Measure: Mean (Standard Deviation); unit: change in percentage of TTR
Arm/Group | Intervention Arm
Number analyzed (Participants) | 50
change in percentage of TTR
  6 months | -12.2 (26.4)
  12 months: number analyzed (Participants) | 49
  12 months | -7.3 (18.3)
  24 months: number analyzed (Participants) | 44
  24 months | -4.4 (13.2)

7. Secondary Outcome: Patient Satisfaction Through Total DASS Score
Description: Patient satisfaction through total DASS score. DASS = Duke Anticoagulation Satisfaction Scale. 25-item scale.Higher numbers indicate worsening satisfaction ranging from 25-175. Seven-point ordinal scale ("not at all" = 1, "very much" = 7).
Time Frame: baseline, 6 months, 12 months, 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 48
score on a scale
  baseline | 42.89 (12.08)
  6 months | 43.99 (11.75)
  12 months | 38.83 (11.53)
  24 months | 46.82 (15.16)

8. Other Pre Specified Outcome: Frequency and Type of Protocol Deviations From Both Participants and Study Staff
Description: This outcome determines the frequency and type of protocol deviations from both participants and study staff
Time Frame: Up to 2.25 years
Population: 634 eligible participant visits
Measure: Number; unit: percentage of visits
Units Other Than Participants: participant visits
Arm/Group | Intervention Arm
Number analyzed (Participants) | 50
Number analyzed (participant visits) | 634
percentage of visits
  extended interval visits scheduled correctly | 94.3
  Deviations too short | 3.0
  Deviations too long | 2.7

ADVERSE EVENTS:
Time Frame: 24 months
Description: Major bleeding was defined as a fatal or symptomatic bleed into a critical area or organ, bleeding leading to hospitalization, or transfusion of two units or more of packed red blood cells. This definition is the standard definition used by the Anticoagulation Clinic to report events.
  Serious bleeding was defined as bleeding leading to emergency or urgent care visit or additional testing required.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 15/50
Other Adverse Events (participants affected / at risk) | 19/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=50)
Multiple myeloma (Blood and lymphatic system disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (2)
Heart failure (Cardiac disorders) | 3 (5)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Severe AKI (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RLE cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
Post-op monitoring for vascular procedure (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=50)
Thromboembolism (Vascular disorders) | 1 (2)
Major bleeding (Blood and lymphatic system disorders) | 6 (6)
Serious bleeding (Blood and lymphatic system disorders) | 16 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT02392104/Prot_SAP_000.pdf